CLINICAL TRIAL: NCT00941408
Title: Biomarker Study of Breast Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: BR03/17/08
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Breast Tumors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — During the diagnostic tumor core biopsy, 3-4 additional tumor samples will be obtained through the same needle track for the purpose of this study. The tumor cores will be stored in liquid nitrogen for subsequent histopathological analysis; DNA, RNA and protein will be extracted from tumor cores for genetic, gene expression and proteomics studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic tumor core biopsy
  Interventions: Procedure: Diagnostic tumor core biopsy

INTERVENTIONS:
Procedure: Diagnostic tumor core biopsy

SUMMARY:
This protocol aims to create a tissue bank of breast tumors obtained at the time of diagnosis for the identification of biomarkers for diagnosis, prognostication, and prediction of treatment response in breast cancer. While tissue banks now exist in major hospitals in Singapore to collect tumor specimens at the time of surgery, specimens collected at surgery from patients who had undergone pre-operative treatment represent a post-treatment sample and not a baseline, untreated sample. Such samples are intrinsically different from untreated samples, and have to be analyzed separately from untreated samples. However, they remain valuable samples, particularly if a pre-treatment sample has been obtained, providing paired pre- and post-treatment samples, which could provide valuable information on treatment-related tumor biomarker changes. A tissue bank comprising of samples collected during the diagnostic core biopsy thus represents a valuable supplement to existing tissue banks.

Approximately 10-20% of patients diagnosed with non-metastatic breast cancer will require neoadjuvant chemotherapy. In addition, future clinical trials may include 'window-of-opportunity' studies during which biological therapy is administered for a short period (2-3 weeks) while an operable breast cancer patient is awaiting definitive surgery. The majority of early-stage breast cancer patients would be eligible for such trials, allowing the rapid recruitment of breast cancer patients. When coupled with analysis of surrogate markers of response (eg apoptosis, anti-angiogenic effects, etc), these unique clinical trials could provide valuable insights into the biological effects of new therapeutic agents in evaluation.

DETAILED DESCRIPTION:
Abstract of Research Proposal:

Breast cancer is a heterogeneous disease, with various subtypes demonstrating differing biological behavior, prognosis, and response to therapeutic agents. Improving the understanding of the biology of breast cancer can result in better prognostication and therapy in individual patients, and has important clinical implications. While valuable scientific knowledge is generated from studies of breast cancer cell lines or animal models, such information generated in vitro may not fully reflect the in vivo model. Direct analysis of patient samples is important to validate in vitro findings, and represents a step closer to clinical application. Studying patient tumor samples for genetic and protein markers and correlating these analyses with clinical characteristics and outcomes could provide valuable insights into tumor biology in vivo, and leads to better understanding of tumor biology and resistance mechanisms. This is a single-centre study of biomarker analysis in breast tumors. A total of 400 patients with breast lesions for whom a diagnostic core biopsy is planned will be enrolled over 2 years. During the diagnostic tumor core biopsy, 3-4 additional tumor samples will be obtained through the same needle track for the purpose of this study. The tumor cores will be stored in liquid nitrogen for subsequent histopathological analysis; DNA, RNA and protein will be extracted from tumor cores for genetic, gene expression and proteomics studies. The patient's clinical progress will be tracked through the clinical case files. For patients in whom the clinical diagnostic biopsy yields a benign result, the samples obtained from them will serve as control specimens. For patients in whom the clinical diagnostic core biopsy confirms the diagnosis of breast cancer, the samples will be considered cases, and the following information will be tracked: histopathological characteristics of the tumor including ER/PR/c-erbB2 status and other known prognostic and predictive immunohistochemical markers (e.g., Ki67, p53, etc), anti-cancer treatment, progression-free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Suspicious breast lesion for which diagnostic core biopsy is planned.
* Patients must not have received prior or scheduled to receive chemotherapy, hormonal therapy, radiotherapy, targeted therapy, or immunotherapy for the treatment of breast cancer.
* Signed informed consent from patient or legal representative.

Exclusion Criteria:

* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast lesions for whom a diagnostic core biopsy is planned
Sampling Method: Non-Probability Sample
Enrollment: 400
Dates: Start 2009-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Mouridsen HT, Andersen AP, Brincker H, Dombernowsky P, Rose C, Andersen KW. Adjuvant tamoxifen in postmenopausal high-risk breast cancer patients: present status of Danish Breast Cancer Cooperative Group trials. NCI Monogr. 1986;(1):115-8. PMID 3534583
- [Background] Gaskell DJ, Hawkins RA, Sangsterl K, Chetty U, Forrest AP. Relation between immunocytochemical estimation of oestrogen receptor in elderly patients with primary breast cancer and response to tamoxifen. Lancet. 1989 May 13;1(8646):1044-6. doi: 10.1016/s0140-6736(89)92445-8. PMID 2566000